CLINICAL TRIAL: NCT06419933
Title: Prevention of Emotional Problems in Preschool Children Aged to 4 to 6 Years Old: Evaluation of the SuperKids Program (PRE-KIDS)
Brief Title: Emotional Problems in Preschool Children: Evaluation of the SuperKids Program (PRE-KIDS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Mireia Orgilés Amorós, professor, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PID2021-126473NB-I00
Record Dates: First submitted 2024-05-08; First posted 2024-05-17 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-05

CONDITIONS: Emotional Problem
Keywords: Social skills; Emotional skills; Program evaluation; Preschool children
MeSH Terms: conditions — Social Skills

STUDY DESIGN:
Intervention Model Description: Cross-assignment. Participants who meet the inclusion criteria and undergo the full baseline assessment will be assigned to the intervention group condition or to the WLC group. Children assigned to the intervention condition will receive the eight-week intervention. Participants in the WLC group will not receive any psychological intervention during the eight-week program. Children and parents in all groups will complete the same set of measures at approximately the same time (pre-test and post-eight weeks). Children in the WLC group will receive the intervention after the follow-up visit is completed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group wait-list (No Intervention): Group without any intervention. Participants in the wait-list group will receive no psychological intervention during the eight-week duration of the SuperKids program. Families will be informed that children in this group will receive the intervention once the follow-up is completed.
- Experimental group (Experimental): SuperKids Structured and manualized intervention with a manual for the therapist and a workbook for the children. The intervention will be administered by SuperKids-trained clinical psychologists. Sessions will take place once a week for eight weeks, with each session lasting approximately forty-five minutes. The program includes emotional education and social skills training. These contents are learned through playful exercises, activities, readings and role-playing. The intervention modality will be face-to-face.
  Interventions: Other: The SuperKids Program

INTERVENTIONS:
Other: The SuperKids Program — The SuperKids program will be administered following the manual of the intervention by a trained therapist, as described in the section of intervention/ treatment
  Arms: Experimental group

SUMMARY:
Emotional problems are among the most frequent psychological problems in the school stage, having an early onset. When they are not detected and they do not receive adequate intervention, they persist and become chronic, being considered precursors of other problems in adolescence and adulthood. The early onset of emotional problems, and their precursor role for other disorders, justify the need for preventive interventions as soon as possible. Since there is evidence that anxiety and depression share common underlying mechanisms, preventive programs should address shared risk factors. For this reason, the objective of this study is to test the effectiveness of an 8-session cognitive-behavioral protocol developed for Spanish children aged 4 to 6 in the educational context in a controlled trial. The objective of the program is that children improve their skills to manage their own emotions and to improve their ability to interact with other. The program will be applied ina group format and will be enriched with multimedia material that the implementer will project at various moments of the sessions.

DETAILED DESCRIPTION:
A 2 x 3 factorial design will be used, with the intervention variable as an intergroup factor (intervention or waiting list), and with the evaluation phase as an intragroup factor (pretest, posttest, 12 months follow-up). Parents and children will complete the same measures at baseline, post-treatment, and follow-up. The investigators will compare the results of pre- and post-assessments of children participating in the program on emotional and social variables.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 6 years.

Exclusion Criteria:

* Intellectual disability, behavioral symptoms or autistic spectrum symptoms whose severity prevented the continuation of treatment.
* Current psychological or pharmacological treatment for anxiety and/or depression.
* Not accepting or revoking informed consent to participate in the study.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The Kiddy-KINDL-R | Before starting the study
  Baseline level of physical and emotional well-being reported by parents as measured by the Kiddy-KINDL-R questionnaire. The Kiddy-KINDL-R measures assesses physical and emotional well-being of children aged 4 to 7 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Parents rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate higher symptoms in children.
The Kiddy-KINDL-R | Immediately after the intervention.
  Level of physical and emotional well-being reported by parents immediately after the intervention measured by the Kiddy-KINDL-R questionnaire. The Kiddy-KINDL-R measures assesses physical and emotional well-being of children aged 4 to 7 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Parents rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate higher symptoms in children.
The Kiddy-KINDL-R | 12 months after the intervention.
  Level of physical and emotional well-being reported by parents at 12 months Measured by the Kiddy-KINDL-R questionnaire. The Kiddy-KINDL-R measures assesses physical and emotional well-being of children aged 4 to 7 years across six dimensions: physical well-being, psychological well-being, self-esteem, family, social relationships, and school. Parents rate each item on a 5-point Likert scale: never (1), almost never (2), sometimes (3), almost always (4), and always (5). The total score is calculated by adding the scores for each dimension (range for each dimension: 4 to 20 points). Higher scores on each subscale and on the total scale indicate higher symptoms in children.
Preschool Spence Anxiety Scale (PAS) | Before starting the study
  Baseline child-reported anxiety symptoms as measured by the Preschool Spence Anxiety Scale (PAS). The PAS measures symptom severity of DSMIV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety, and specific fears). The frequency of symptoms is recorded on a 3-point Likert scale from 0 (never) to 3 (always). A minimum possible score of 0 and a maximum possible score of 114 is obtained. Higher scores indicate greater symptom severity. Higher scores indicate greater symptom severity.
Preschool Spence Anxiety Scale (PAS) | Immediately after the intervention.
  Anxiety symptoms reported by children immediately after the intervention measured using the Spence Preschool Anxiety Scale, (PAS). The PAS measures symptom severity of DSMIV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety, and specific fears). The frequency of symptoms is recorded on a 3-point Likert scale from 0 (never) to 3 (always). A minimum possible score of 0 and a maximum possible score of 114 is obtained. Higher scores indicate greater symptom severity. Higher scores indicate greater symptom severity.
Preschool Spence Anxiety Scale (PAS) | 12 months after the intervention.
  Child-reported anxiety symptoms at 12 months Measured using the Spence Preschool Anxiety Scale (PAS). The PAS measures symptom severity of DSMIV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety, and specific fears). The frequency of symptoms is recorded on a 3-point Likert scale from 0 (never) to 3 (always). A minimum possible score of 0 and a maximum possible score of 114 is obtained. Higher scores indicate greater symptom severity. Higher scores indicate greater severity of symptoms.
the Strengths and Difficulties Questionnaire | Before starting the study
  Baseline Parent-reported depressive symptoms as measured by the Strengths and Difficulties Questionnaire, parent version (SDQ; Goodman, 1997). The SDQ measure examines emotional difficulties (5 items), conduct problems (5 items), hyperactivity (5 items), peer problems (5 items), and prosocial behavior (5 items) in children aged 3 to 16 years. Symptom frequency is recorded on a 3-point Likert scale from 0 (Not true) to 3 (Absolutely true). A minimum possible score of 0 and a maximum possible score of 114 is obtained. Higher scores indicate greater severity of symptoms. Higher scores indicate greater symptom severity.
the Strengths and Difficulties Questionnaire | Immediately after the intervention.
  Depressive symptoms reported by parents inmediately after intervention measured by the Strengths and Difficulties Questionnaire, parent version (SDQ; Goodman, 1997). The SDQ measure examines emotional difficulties (5 items), conduct problems (5 items), hyperactivity (5 items), peer problems (5 items), and prosocial behavior (5 items) in children aged 3 to 16 years. Symptom frequency is recorded on a 3-point Likert scale from 0 (Not true) to 3 (Absolutely true). A minimum possible score of 0 and a maximum possible score of 114 is obtained. Higher scores indicate greater severity of symptoms. Higher scores indicate greater symptom severity.
the Strengths and Difficulties Questionnaire | 12 months after the intervention.
  Depressive symptoms reported by parents at 12 months as measured by the Strengths and Difficulties Questionnaire, parent version (SDQ; Goodman, 1997). The SDQ measure examines emotional difficulties (5 items), conduct problems (5 items), hyperactivity (5 items), peer problems (5 items), and prosocial behavior (5 items) in children aged 3 to 16 years. Symptom frequency is recorded on a 3-point Likert scale from 0 (Not true) to 3 (Absolutely true). A minimum possible score of 0 and a maximum possible score of 114 is obtained. Higher scores indicate greater severity of symptoms. Higher scores indicate greater symptom severity.
Behavioral Inhibition Questionnaire (BIQ | Before starting the study
  Baseline of children's behavioral inhibition measured using the Behavioral Inhibition Questionnaire (BIQ). The BIQ assesses the frequency of children's behavioral inhibition in six contexts across three domains: social novelty (unknown adults, peers, and performance in front of others), situational novelty (unfamiliar situations, preschool/separation), and novel physical activities with a possible risk of injury. This questionnaire has 30 items that are scored on a seven-point scale ranging from 1 (almost never) to 7 (almost always). Item scores are summed to create six scale scores: Unknown Peers, Unknown Adults, Performance Situations, Separation/Preschool, Unknown Situations, and Physically Challenging Situations.
Behavioral Inhibition Questionnaire (BIQ | Immediately after the intervention.
  Children's behavioral inhibition was immediately measured after the intervention using the Behavioral Inhibition Questionnaire (BIQ). The BIQ assesses the frequency of children's behavioral inhibition in six contexts across three domains: social novelty (unknown adults, peers, and performance in front of others), situational novelty (unfamiliar situations, preschool/separation), and novel physical activities with a possible risk of injury. This questionnaire has 30 items that are scored on a seven-point scale ranging from 1 (almost never) to 7 (almost always). Item scores are summed to create six scale scores: Unknown Peers, Unknown Adults, Performance Situations, Separation/Preschool, Unknown Situations, and Physically Challenging Situations.
Behavioral Inhibition Questionnaire (BIQ | 12 months after the intervention.
  Children's behavioral inhibition was measured at 12 months using the Behavioral Inhibition Questionnaire (BIQ). The BIQ assesses the frequency of children's behavioral inhibition in six contexts across three domains: social novelty (unknown adults, peers, and performance in front of others), situational novelty (unfamiliar situations, preschool/separation), and novel physical activities with a possible risk of injury. This questionnaire has 30 items that are scored on a seven-point scale ranging from 1 (almost never) to 7 (almost always). Item scores are summed to create six scale scores: Unknown Peers, Unknown Adults, Performance Situations, Separation/Preschool, Unknown Situations, and Physically Challenging Situations.
Parental Overprotection Scale | Baseline
  Parental overprotective behavior is assessed with the Parental Overprotection Scale (OP, Edwards et al., 2008). POM evaluates, through 19 items, the overprotective behavior of parents towards their children, related in previous studies to anxiety in preschool children. Symptom frequency is recorded on a 3-point Likert scale, from 0 (not at all) to 4 (very much).
Depression Anxiety Stress Scales - short version (DASS-21) | Baseline
  Baseline parental depression, anxiety and stress symptoms Measured by the Depression Anxiety Stress Scales - short version (DASS-21). It contains a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic nonspecific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Orgilés Amorós, Principal Investigator — Universidad Miguel Hernandez de Elche
Locations (1):
- Department of Health Psychology. Miguel Hernandez University of Elche Elche, Alicante, Spain, 03202, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bishop G, Spence SH, McDonald C. Can parents and teachers provide a reliable and valid report of behavioral inhibition? Child Dev. 2003 Nov-Dec;74(6):1899-917. doi: 10.1046/j.1467-8624.2003.00645.x. PMID 14669903
- [Background] Orgiles M, Melero S, Penosa P, Espada JP, Morales A. [Parent-reported Health-Related Quality of Life in Spanish pre-schoolers: Psychometric properties of the Kiddy-KINDL-R]. An Pediatr (Engl Ed). 2019 May;90(5):263-271. doi: 10.1016/j.anpedi.2018.04.019. Epub 2018 Jul 6. Spanish. PMID 31056090
- [Background] Orgiles M, Penosa P, Fernandez-Martinez I, Marzo JC, Espada JP. Spanish validation of the Spence Preschool Anxiety Scale. Child Care Health Dev. 2018 Sep;44(5):753-758. doi: 10.1111/cch.12593. Epub 2018 Jul 22. PMID 30033647